CLINICAL TRIAL: NCT01503138
Title: The Effect of a Purpose-built Intervention on Mental Health in Mainland Chinese Immigrant Women Survivors of Intimate Partner Violence: A Randomized Controlled Trial
Brief Title: Intervention for Abused Chinese Immigrant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, TIWARI, Agnes, Professor and Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 11-051
Record Dates: First submitted 2011-12-30; First posted 2012-01-02 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Mental Health Wellness 1; Domestic Violence
Keywords: Intimate Partner Violence; Depressive Symptoms; Intervention; Randomized Controlled Trial; Mainland Chinese; Immigrants; Women
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purpose-built intervention (Experimental): A purpose-built intervention consists of: (i) Empowerment; (ii) Parenting workshops; and (iii) Telephone social support and Peer support.
  Interventions: Behavioral: Purpose-built intervention
- Standard community health education program (No Intervention): The community health education programme consists of two group sessions with one on the topic of osteoporosis and one on dietary therapy based on the concepts of Chinese medicine.

INTERVENTIONS:
Behavioral: Purpose-built intervention — A purpose-built intervention consists of: (i) Empowerment; (ii) Parenting workshops; and (iii) Telephone social support and Peer support.
  Arms: Purpose-built intervention

SUMMARY:
The purpose of this study is to evaluate the efficacy of a purpose-built intervention in improving the mental health of abused Mainland Chinese immigrant women in a community in Hong Kong.

DETAILED DESCRIPTION:
Depression is one of the most common mental health sequelae of Intimate partner violence. Not only does depression have an adverse effect on abused women's health and well-being, it also reduces their capacity to cope with the abuse by limiting their ability to perform self-care, meet work requirement, maintain independence, establish relationships, and access social support. Previously, the ability of abused women to take care of themselves was found to be a protective factor for depression. In order to enhance abused women's self-care, advocacy interventions have been developed to help them make sense of the abusive situation, identify potential solutions, and achieve their goals. Also, immigration status was shown to be significantly associated with a higher level of depressive symptoms among the abused women. The findings are important as they point to the need for further research to develop and evaluate culturally congruent interventions to meet the needs of abused Mainland Chinese immigrant women in Hong Kong. Therefore, the purpose of this study is to develop a purpose-built intervention to address the unmet needs of Mainland Chinese immigrant women survivors of Intimate partner violence and to assess its effect on the mental health of the women.

ELIGIBILITY:
Inclusion Criteria:

* Mainland Chinese immigrant women,
* 18 years of age or older,
* holding a one-way or two-way permit,
* have settled in Hong Kong with their intimate partners for less than seven years,
* have at least one child under 18 years of age,
* residing in the Kwai Chung, Tsuen Wan or Tsing Yi districts, and
* assessed to be abused by an intimate partner, based on the Abuse Assessment Screen.

Exclusion Criteria:

* participated in our positive parenting program or advocacy intervention previously, or
* will not be in Hong Kong during the intervention/standard health education program or the follow-up telephone interview, or
* is abused by someone who is not her intimate partner, or
* is unable to communicate in Cantonese or Putonghua.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms at 6-month post-intervention | Baseline and 6-month post-intervention
  The Beck Depression Inventory version II is used to assess depressive symptoms at baseline and also at 6-month post-intervention

SECONDARY OUTCOMES:
Change from baseline in parenting stress at 6-month post-intervention | Baseline and 6-month post-intervention
  The Parenting Stress Index is used to measure paretning stress at baseline and also at 6-month post-intervention
Change from baseline in perceptions of social support at 6-month post-intervention | Baseline and 6-month post-intervention
  The 12-item Interpersonal Support Evaluation List is used to assess perceptions of social supportat baseline and also at 6-month post-intervention
Change from baseline in health-related quality of life at 6-month post-intervention | Baseline and 6-month post-intervention
  The SF-12 Health Survey is used to assess health-related quality of life at baseline and also at 6-month post-intervention
Change from baseline in intimate partner violence at 6-month post-intervention | Baseline and 6-month post-intervention
  The Revised Conflict Tactics Scales is used to measure the type and frequency of behaviors used by the perpetrator during partner conflict at baseline and also at 6-month post-intervention.
Change from baseline in safety behaviors at 6-month post-intervention | Baseline and 6-month post-intervention.
  The Safety Assessment Checklist is used to to measure the safety behaviours used by abused women to avert intimate partner violence at baseline and also at 6-month post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Tiwari, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- HKSKH Lady MacLehose Center, Hong Kong, China

REFERENCES:
- [Background] Golding JM. Intimate partner violence as a risk factor for mental disorders: a meta-analysis. J Fam Viol 1999; 14: 99-132.
- [Background] Kendall-Tackett KA. Inflammation, cardiovascular disease, and metabolic syndrome as sequelae of violence against women: the role of depression, hostility, and sleep disturbance. Trauma Violence Abuse. 2007 Apr;8(2):117-26. doi: 10.1177/1524838007301161. PMID 17545569
- [Background] Constantino RE, Sekula LK, Rabin B, Stone C. Negative life experiences, depression, and immune function in abused and nonabused women. Biol Res Nurs. 2000 Jan;1(3):190-8. doi: 10.1177/109980040000100304. PMID 11232214
- [Background] Brush LD. Battering, traumatic stress, and welfare-to-work transition. Violence Against Women 2000; 6:1039-1065.
- [Background] O'Brien SM. Staying alive: a client with chronic mental illness in an environment of domestic violence. Holist Nurs Pract. 2002 Apr;16(3):16-23. doi: 10.1097/00004650-200204000-00006. PMID 11913224
- [Background] Carlson BE, McNutt L, Choi DY, Rose IM. Intimate partner abuse and mental health: The role of social support and other protective factors. Violence Against Women 2002; 8: 720-745.
- [Background] Campbell JC, Kub J, Belknap RA, Templin TN. Predictors of depression in battered women. Violence Against Women 1997; 3: 271-93. PMID: 12349116
- [Background] Ford-Gilboe M, Varcoe C, Wuest J, Merritt-Gray M. Intimate partner violence and nursing practice. In Humphreys J, Campbell JC, eds. Family violence and nursing practice (2nd ed). New York: Springer 2010; 115-154.
- [Background] Wong JY, Tiwari A, Fong DY, Humphreys J, Bullock L. Depression among women experiencing intimate partner violence in a Chinese community. Nurs Res. 2011 Jan-Feb;60(1):58-65. doi: 10.1097/NNR.0b013e3182002a7c. PMID 21127447